CLINICAL TRIAL: NCT06972823
Title: Assessing Changes in Oral Functions and Speech After Using 3D-Printed vs. Custom-made Mouth Guards in Children Practicing Contact Sports: A Randomized Clinical Trial
Brief Title: Impact of 3D-Printed and Custom Mouthguards on Speech and Oral Functions in Children Practicing Contact Sports
Acronym: Mouthguards
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yasir mohammed hassan aljadani, Master's Candidate, Department of Pediatric Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Custom Mouthguards and Speech
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Mouthguard Use; Orofacial Injuries Prevention; 3D Printed Mouthguard; Traditional Custom-made Mouthguard; Speech and Oral Functions
Keywords: 3D printed mouthguard; traditional custom-made mouthguard; speech; oral functiions; CAD/CAM; 3D printer; Children; Pediatric Dentistry; Contact sports; speaking
MeSH Terms: conditions — Speech

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two groups: one group will receive traditional custom-made mouthguards, and the other will receive 3D-printed custom-made mouthguards. Each participant will remain in their assigned group throughout the study period, and outcomes will be assessed independently for each group.
Who Masked: Participant, Investigator
Masking Description: Blinding will be applied at multiple levels to minimize bias in this study. Since both the traditional custom-made and 3D-printed mouthguards have a similar appearance, this study will be double-blinded to both the principal investigator and the patients in each study group, thereby reducing expectation bias. A coach, who is not involved in data collection or analysis, will be responsible for distributing the mouthguards to participants, ensuring that neither the principal investigator nor the participants know which type of mouthguard is being used. Additionally, the assessors evaluating speech and oral function will remain blinded to the type of mouthguard. To further ensure objective data analysis and minimize detection and reporting bias, the statistician will also be fully blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed custom-made mouthguards (Experimental): This arm will include participants receiving 3D printed custom mouthguards.
  Interventions: Device: 3D printed custom-made mouthguards
- Traditional custom-made mouthguards (Active Comparator): Participants in the second group will receive traditional custom-made mouthguards.
  Interventions: Device: Traditional custom-made mouthguards

INTERVENTIONS:
Device: 3D printed custom-made mouthguards — Participants in the first group will receive 3D printed custom-made mouthguards
  Arms: 3D printed custom-made mouthguards
Device: Traditional custom-made mouthguards — Participants in the active comparator arm will receive traditional custom-made mouthguards as an intervention
  Arms: Traditional custom-made mouthguards

SUMMARY:
This study aims to compare the effects of traditional and 3D-printed custom-made mouthguards on speech and oral functions in pediatric cases who practice contact sports by evaluating the comfort, fit, and performance of both types of mouthguard fabrication methods. The study will be conducted on 60 children who practice contact sports, and the changes in speech, oral functions, the occlusal thickness of the mouthguards, and the cost efficiency will be assessed over a period of one year.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at Cairo International Stadium, enrolling healthy children aged 8 to 14 who are actively engaged in contact sports and require mouthguards for protection. Eligible participants must be cooperative and have no history of speech or neurological disorders, orthodontic treatment, or dental anomalies that may affect mouthguard adaptation. After obtaining informed consent from parents, participants will be randomly allocated in a 1:1 ratio into two groups.

Group 1 will receive traditional custom-made mouthguards fabricated from alginate impression material. Group 2 will receive 3D-printed custom-made mouthguards created from digital intraoral scans using CAD/CAM and 3D printing technology. All fittings will be adjusted for comfort, retention, and occlusal balance by the principal investigator.

The primary outcomes include changes in oral functions and speech, assessed using a validated Likert-scale questionnaire adapted from Mat Zainal et al. (2024), administered at baseline, 3 months, and 6 months. Secondary outcomes include evaluating the knowledge, attitude, and practice (KAP) toward mouthguard use using a structured questionnaire (Vignesh et al., 2023), cost efficiency via the incremental cost-effectiveness ratio (ICER), and occlusal thickness changes using an Iwanson caliper. This trial aims to determine whether 3D-printed mouthguards provide superior or equivalent function, comfort, and cost-efficiency compared to traditional methods, potentially advancing the standards of pediatric sports dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-14 years of both ages.
* Participants actively engaged in contact sports.
* Children who require mouthguards for protection.
* Cooperative children.

Exclusion Criteria:

* Children with a history of speech or neurological disorders affecting oral function
* Parental refusal to participate.
* Children currently undergoing orthodontic treatment with fixed appliances.
* Presence of severe dental anomalies or extensive missing teeth that could interfere with mouthguard adaptation.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Changes Speech and in Oral Functions | Six months
  Oral functions, including speaking difficulty, lisping, nausea, bulkiness, and mouth dryness, will be assessed using a validated questionnaire adapted from the study by Mat Zainal et al. (2024). The questionnaire will be administered at three distinct intervals (baseline, 3 months, and six months)

SECONDARY OUTCOMES:
Knowledge, attitude, and practice (KAP) of children toward mouthguards | initial visit (the first month)
  The study will evaluate the knowledge, attitudes, and practices (KAP) of children regarding the use of mouthguards in preventing orofacial injuries during contact sports. Specifically, the study assesses children's awareness of the risks of orofacial injuries, their understanding of mouthguards as a protective measure, and their current usage patterns. Based on a previous study by Vignesh et al. (2023), a structured and well-adapted questionnaire will be given to all participants in both groups at the initial visit.
Cost Efficiency of both mouthguards | one year
  This study will also assess the cost efficiency of both types of custom-made mouthguards by calculating the cost per unit, using the U.S Dollar (USD) as the unit of measurement. The incremental cost effectiveness ratio will be calculated after one year.
  The following equation will be used to measure the incremental cost-effectiveness ratio (Sadatsafavi et al., 2009):
  ICER=(Mouthguard A cost- Mouthguard B cost)/(outcome of mouthguard A-Outcome of mouthguard B)
Occlusal thickness changes | Three months
  This study will assess the wear patterns of both types of mouthguards in children participating in contact sports. The wear patterns will be measured by evaluating the thickness reduction of the mouthguards over time using an Iwanson caliper (measured in millimeters, mm). This method will provide quantitative data on the durability and wear resistance of each type of mouthguard, helping to determine which type maintains its protective properties longer under the stress of regular use (Tewari et al., 2024). The mouthguard thickness will be measured at two distinct timepoints (baseline and three months)

CONTACTS AND LOCATIONS:
Overall Officials: Gihan M Abuelniel, Doctoral Degree (Professor), Study Director — Cairo University; Passant Nagi, Master's Degree, Study Director — Cairo University
Locations (1):
- Faculy of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be shared with qualified researchers upon request, following ethical guidelines and approval from the relevant ethics committee. The data will be anonymized to ensure participant confidentiality and will be made available through a secure data repository.

REFERENCES:
- [Background] Vignesh, T. S., Chinni, S. K., Anumula, L., Sannapureddy, S., Kumar, Y. P., & Rohith, V. V. S. (2023). Knowledge, Attitudes, and Practices of Mouth Guards in the Prevention of Orofacial Injuries in Sports Persons-A Cross-sectional Study. Journal of Interdisciplinary Dentistry, 13(2), 84-89.
- [Background] Tewari N, Kahler B, Srivastav S, Goel S. How far have we come? A historic scoping review of dental traumatology literature. Dent Traumatol. 2022 Oct;38(5):345-355. doi: 10.1111/edt.12760. Epub 2022 May 25. PMID 35612349
- [Background] Tanaka Y, Maeda Y, Yang TC, Ando T, Tauchi Y, Miyanaga H. Prevention of orofacial injury via the use of mouthguards among young male rugby players. Int J Sports Med. 2015 Mar;36(3):254-61. doi: 10.1055/s-0034-1390498. Epub 2014 Oct 20. PMID 25329428
- [Background] Sousa AM, Pinho AC, Messias A, Piedade AP. Present Status in Polymeric Mouthguards. A Future Area for Additive Manufacturing? Polymers (Basel). 2020 Jul 3;12(7):1490. doi: 10.3390/polym12071490. PMID 32635307
- [Background] Singh G, Garg S, Damle SG, Dhindsa A, Kaur A, Singla S. A study of sports related occurrence of traumatic orodental injuries and associated risk factors in high school students in north India. Asian J Sports Med. 2014 Sep;5(3):e22766. doi: 10.5812/asjsm.22766. Epub 2014 Aug 28. PMID 25520762
- [Background] Sadatsafavi M, Marra CA, Ayas NT, Stradling J, Fleetham J. Cost-effectiveness of oral appliances in the treatment of obstructive sleep apnoea-hypopnoea. Sleep Breath. 2009 Aug;13(3):241-52. doi: 10.1007/s11325-009-0248-4. Epub 2009 Feb 20. PMID 19229577
- [Background] Roberts HW. Sports mouthguard overview: Materials, fabrication techniques, existing standards, and future research needs. Dent Traumatol. 2023 Apr;39(2):101-108. doi: 10.1111/edt.12809. Epub 2022 Nov 27. PMID 36436198
- [Background] Ntovas P, Ladia O, Kois JC, Rahiotis C, Revilla-Leon M. Digital workflow for the fabrication of custom-fit additively manufactured sports mouthguards with balanced occlusion using an optical jaw tracking system: A dental technique. J Prosthet Dent. 2025 Nov;134(5):1536-1541. doi: 10.1016/j.prosdent.2024.07.021. Epub 2024 Aug 22. PMID 39174379
- [Background] Mordini L, Lee P, Lazaro R, Biagi R, Giannetti L. Sport and Dental Traumatology: Surgical Solutions and Prevention. Dent J (Basel). 2021 Mar 23;9(3):33. doi: 10.3390/dj9030033. PMID 33806915
- [Background] Mat Zainal MK, Liew AKC, Abdullah D, Soo E, Abdul Hamid B, Ramlee RAM. Changes in oral functions and speech when using custom-fitted mouthguards: An uncontrolled before-and-after study. Dent Traumatol. 2024 Aug;40(4):460-469. doi: 10.1111/edt.12939. Epub 2024 Mar 8. PMID 38459669
- [Background] Green JI. The Role of Mouthguards in Preventing and Reducing Sports-related Trauma. Prim Dent J. 2017 May 1;6(2):27-34. doi: 10.1308/205016817821281738. PMID 28668098
- [Background] Dias Goncalves VP, Fontes Vieira CM, Colorado Lopera HA. The production and materials of mouthguards: Conventional vs additive manufacturing - A systematic review. Heliyon. 2024 Jul 8;10(14):e34294. doi: 10.1016/j.heliyon.2024.e34294. eCollection 2024 Jul 30. PMID 39092246
- [Background] Dolic O, Obradovic M, Kojic Z, Knezevic N, Trtic N, Veselinovic V, Arapovic-Savic M, Umicevic-Davidovic M, Krcic V. Traumatic Dental Injuries in Children and Adolescents from a Major Dental Clinic in Bosnia and Herzegovina: A 5-Year Retrospective Study. Medicina (Kaunas). 2024 Nov 8;60(11):1843. doi: 10.3390/medicina60111843. PMID 39597028
- [Background] Del Rossi G, Lisman P, Signorile J. Fabricating a better mouthguard. Part II: the effect of color on adaptation and fit. Dent Traumatol. 2008 Apr;24(2):197-200. doi: 10.1111/j.1600-9657.2007.00570.x. PMID 18352924
- [Background] De Queiroz, T. S., da Cruz, B. S., Demachkia, A. M. M., Borges, A. L. S., Tribst, J. P. M., & Paes Junior, T. J. d. A. (2023). Ergonomic sports mouthguards: A narrative literature review and future perspectives. Applied Sciences, 13(20), 11353.
- [Background] Borin-Moura, L., Azambuja-Carvalho, P., Daer-de-Faria, G., Barros-Gonçalves, L., Kirst-Post, L., & Braga-Xavier, C. (2018). A 10-year retrospective study of dental trauma in permanent dentition. Revista Española de Cirugía Oral y Maxilofacial, 40(2), 65-70.
- [Background] Avgerinos S, Stamos A, Nanussi A, Engels-Deutsch M, Cantamessa S, Dartevelle JL, Unamuno E, Del Grosso F, Fritsch T, Crouzette T, Striegel M, Sanchez CC, Okshah A, Tzimpoulas N, Naka O, Kouveliotis G, Tzoutzas I, Zoidis P, Synodinos F, Loizos E, Tasopoulos T, Haughey J, Rahiotis C. Position Statement and Recommendations for Custom-Made Sport Mouthguards. Dent Traumatol. 2025 Jun;41(3):246-251. doi: 10.1111/edt.13019. Epub 2024 Nov 22. PMID 39578680
- [Background] Abbott PV, Tewari N, Mills SC, Stasiuk H, Roettger M, O'Connell AC, Levin L. The International Association of Dental Traumatology (IADT) and the Academy for Sports Dentistry (ASD) guidelines for prevention of traumatic dental injuries: Part 4: Faceshields for the prevention of dental and oral trauma. Dent Traumatol. 2024 Feb;40 Suppl 1:10-11. doi: 10.1111/edt.12926. PMID 38363703
- See also: Related Info — https://www.researchgate.net/publication/383066550_3D_Printed_customized_sports_mouthguard